CLINICAL TRIAL: NCT05985083
Title: A Phase I, Open-Label, Multicenter, Dose-Escalation And Cohort-Expansion Study Of IMM47 In Subjects With Advanced Solid Tumors
Brief Title: A Study Of IMM47 In Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Collaborators: IQVIA RDS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMM47-201
Record Dates: First submitted 2023-07-30; First posted 2023-08-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Oncology
Keywords: ADVANCED SOLID TUMORS
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation (Experimental): It's a dose escalation to identify the Maximum Tolerated dose (MTD) , recommended Phase II dose (RP2D) of IMM47, an accelerated titration method and the traditional "3+3" design method will be adopted. IMM47 will be sequentially escalated at the dose of 5 μg/kg，50 μg/kg, 250 μg/kg，1.0 mg/kg，3.0 mg/kg and 5.0 mg/kg or higher dose levels, administered via intravenous infusion every 2 weeks in 28-day treatment cycles.
  The duration of the infusion is 120 min (± 10 min) for the 1st infusion and 60 min (± 5 min) for subsequent infusions.
  Interventions: Drug: IMM47

INTERVENTIONS:
Drug: IMM47 — IMM47 is humanized mAb targeting CD24 to be administered via intravenous infusion every 2 weeks in 28-day treatment cycles.

SUMMARY:
This is a first-in-human (FIH), open-label, multi-center, phase I study to evaluate the safety, tolerance, pharmacokinetics (PK), immunogenicity, preliminary anti-tumor activity, pharmacodynamics, and biomarker activity of IMM47 monotherapy in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
In phase Ia phase, approximately 17-48 eligible subjects with advanced solid tumors will be enrolled, and an accelerated titration method and the traditional "3+3" design method will be adopted to explore the safety, tolerability, PK, immunogenicity, and anti-tumor activity of 6 dose levels of IMM47: 5 μg/kg, 50 μg/kg, 250 μg/kg, 1.0 mg/kg, 3.0 mg/kg and 5.0 mg/kg or higher, to determine the MTD and RP2D.

Accelerated dose cohorts: At the dose cohorts of 5 μg/kg and 50 μg/kg, one subject will be enrolled at first, and the conventional "3+3" design will be altered and the additional 2 or 5 subjects would be enrolled if any ≥ Grade 2 drug related toxicities are observed during the first 28-day cycle (DLT observational period).

"3+3" dose cohorts: Thereafter, at least three subjects will be enrolled in each dose cohort at the 250 μg/kg, 1.0 mg/kg, 3.0 mg/kg and 5.0 mg/kg dose levels sequentially. There will be a minimum interval of 48 hours between the 1st and 2nd subjects being dosed in each "3+3" dose cohort. If no DLTs occur in a dose cohort of 3 subjects during the first cycle (DLT observational period), 3 subjects will be enrolled at the next higher dose level. If 1 of 3 subjects in a cohort experiences a DLT, an additional 3 subjects will be enrolled at that dose level. If only 1 of 6 subjects experiences a DLT, then 3 subjects will be enrolled at the next higher dose level. If 2 or more subjects experienced DLTs within a cohort, dose escalation will be halted and 3 more subjects will be enrolled at the previous lower (tolerated) dose level until that cohort has 6 evaluable subjects. Depending on toxicity, the dose deescalation to an intermediate dose may occur. Higher doses than 5.0 mg/kg may be explored under the decision of Safety Review Committee (SRC). A total of 6 subjects must be enrolled at the MTD (or the highest dose studied where no more than 1 of 6 subjects experiences a DLT if the MTD is not identified) and evaluated at the end of Cycle 1 before any subject is dosed in the expansion cohorts.

Continued dosing with IMM47 beyond the second cycle will be offered to subjects who do not experience disease progression or significant toxicity. Subjects who are benefiting from IMM47 will receive the treatment up to 12 cycles, at investigator's discretion. Subjects discontinuing the study treatment early for any reason will complete an end-of-treatment (EOT) visit within 30 (+7) days after the last dose, and a safety follow-up visit within 90 (±7) days after the last dose. If the subjects who achieve complete response (CR), partial response (PR), or stable disease (SD) with clinical benefit discontinue the investigational product, the follow-up visits will be completed every 12 weeks until disease progression, informed consent withdrawn by subject, death, or loss to follow-up, or end of study (whichever occurs first). Survival follow-up will be performed for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the ICF.
2. With an expected life expectancy of ≥ 12 weeks.
3. With an ECOG performance status score of 0-1.
4. For phase Ia, subjects diagnosed histologically or cytologically with advanced solidtumors (preferred but not limited to ovarian, esophageal, breast, lung, colorectal, hepatocellular, pancreatic, urothelial, prostate, and head and neck cancers) that have failed previous standard treatments or no standard treatment is available.
5. The intervals for discontinuing the last anti-tumor therapy prior to the first dose of the investigational product are required as follows Subjects who previously received chemotherapeutic agents must have discontinued the drug for more than 3 weeks.

   Subjects who previously received small-molecule targeted therapy must have discontinued treatment for more than 2 weeks or 5 half-lives of the drug (whichever is longer).

   Subjects who previously received monoclonal antibodies (eg. CD20 antibody, PD-1/PD-L1 antibody) must have discontinued the treatment for more than 4 weeks.

   Subjects who previously underwent palliative radiation therapy must have discontinued the treatment for more than 2 weeks.
6. With suitable organ and hematopoietic functions:

   Neutrophil count ≥1.5 × 109/L. (no growth factor therapy within 4 weeks prior to Screening).

   Platelet count ≥100 × 109/L ; for subjects with HCC, platelet count ≥75 ×109 /L Hemoglobin ≥ 90 g/L (subjects may be transfused >2 weeks before screening, but should not be transfusion-dependent).

   Total Bilirubin (TBIL) ≤ 1.5 × ULN (or ≤ 3.0 × ULN if subject has a documented history of Gilbert's syndrome or liver metastases).

   Both aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN (or both AST and ALT ≤ 5.0 × ULN if subject has a documented history of liver metastases).

   International normalized ratio (INR) ≤1.5 × ULN, or activated partial thromboplastin time (APTT) ≤ 1.5× ULN.

   Left ventricular ejection fraction (LVEF) ≥ 50%. Serum creatinine ≤1.5 × ULN or creatinine clearance (CrCl) ≥ 40 mL/min (Cockcroft and Gault Equation) if serum creatinine >1.5 ULN. Lower calculated creatinine clearance values may be allowed at the Investigator's discretion and in consultation with the Medical Monitor and Sponsor
7. Adverse events associated with previous anti-tumor therapies should have recovered to ≤ Grade 1 (CTCAE version 5.0) (except for toxicities not considered a safety risk such as alopecia, skin pigmentation, and other non-clinically significant abnormalities).
8. Female subjects (based on sex assigned at birth) of childbearing potential must be tested negative for serum pregnancy test during the screening period before receiving the first administration of IMM47; any female subject of childbearing potential must agree to take effective contraceptive measures during the entire study and within 6 months after last dose of the investigational product. A subject is considered to have childbearing potential if he/she is biologically capable of having children and has a heterosexual sex life. Female subjects meeting at least one of the following criteria are deemed to be without childbearing potential:

   Has undergone hysterectomy or bilateral oophorectomy Medically confirmed with ovarian failure Medically confirmed as postmenopausal (menstruation has stopped for 12 consecutive months not for pathological or physiological reasons)

   Acceptable forms of contraception for female subjects are:

   Should not have sexual intercourse or genital contact with a male partner, or use a method of birth control for the duration of the study participation and for 6 months last dose of the investigational product.

   Must agree to use one form of contraception, including sterilization, combined estrogen and progestogen containing hormonal contraception pills or an intravaginal, transdermal, or intrauterine device.

   Intrauterine hormone-releasing system. Bilateral tubal occlusion (surgical procedure that involves blocking by cutting, burning or removing sections, or placing clips of the fallopian tubes to prevent the ovum [egg] from being fertilized).

   A vasectomized partner (surgical procedure that involves cutting and sealing the tubes used to transport semen from the testicles to the penis, thereby rendering infertility).

   Male subjects with female partners of childbearing potential are eligible to participate if they agree to ONE of the following for the duration of the study and until 90 days after the last dose of the study treatment:

   Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

   Agree to use a male condom and have their partner use a contraceptive method with a failure rate of <1% per year as described below when having penile-vaginal intercourse with a WOCBP who is not currently pregnant.

   In addition, male subjects must refrain from donating sperm for the duration of the study and for 90 days after the last dose of study treatment.

   Male subjects with a pregnant or breastfeeding partner must agree to remain abstinent from penile-vaginal intercourse or use a male condom during each episode of penile penetration for the duration of the study and until 90 days after the last dose of the study treatment.
9. Subjects who voluntarily sign the informed consent form, understand the study, and are willing to comply with the protocol, and are able to complete all trial procedures.
10. At least one measurable or evaluable tumor lesion. For solid tumor: Measurable lesion according to RECIST version 1.1 is defined as tumor lesions ≥10 mm in longest diameter or pathologic node ≥ 15 mm in short axis.
11. For both phase Ia and Ib, subjects must agree to provide archived tumor tissue samples for CD24 IHC expression assessment by the central laboratory. In the setting where archival material is unavailable or unsuitable for use (e.g., recently diagnosed subjects or diagnosed with fine needle aspiration), the subject must consent and undergo fresh tumor biopsy (biopsy at acceptable risk as judged by the Investigator). The requirement for fresh biopsy collected from a given subject could be waived after the discussion with the Sponsor, if the tumor tissues are not safely accessible as determined by the Investigator, or the tumor biopsies have to be obtained from sites that require significant risk procedures.

Exclusion Criteria:

1. Subjects who previously received CD24 targeted therapy.
2. Prior allogeneic hematopoietic stem cell transplant or other organ transplants.
3. Subjects with known active central nervous system (CNS) metastases or primary CNS Lymphoma. Stable previously treated CNS metastases in subjects who are asymptomatic and have not been on corticosteroid therapy within 3 weeks prior to screening are not considered to be active.
4. Subjects in need of immediate cytoreduction therapy.
5. Significant medical disease or conditions, as assessed by the Investigators and Sponsor that would substantially increase the risk-benefit ratio of participating in the study. This includes but is not limited to:

   Uncontrolled hypertension (systolic BP > 160 mmHg or diastolic BP > 90 mmHg), pulmonary hypertension, or unstable angina.

   New York Heart Association (NYHA) Grade II or higher congestive heart failure. History of myocardial infarction, or bypass surgery or stent placement within 6 months prior to the first dose of the investigational product.

   Severe arrhythmia requiring treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia that, according to the judgment of the investigators, do not affect the study).

   QTc interval > 450 ms for males and > 470 ms for females (Fridericia's Formula).

   History of cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to the first dose of investigational product.

   Concurrent interstitial lung disease (ILD) (except for radiation therapy-induced loco regional interstitial pneumonia), severe chronic obstructive pulmonary disease, severe pulmonary insufficiency.

   Diseases that may cause gastrointestinal bleeding or perforation. Known inherited or acquired bleeding disorders Uncontrolled diabetes mellitus. Thoracoabdominal or pericardial effusions that cannot be controlled by puncture and drainage and require repeated drainage or with significant symptoms.

   History of liver disease, including cirrhosis, alcoholic liver disease, etc.
6. Concurrent medical condition requiring systemic corticosteroids (prednisone daily dose > 10 mg or equivalent dose) within 7 days prior to first dose of the investigational product or during the study, or other immunosuppressive medications, but not including locoregional corticoids by intranasal, inhalated or other routes of administration, or physiological-dose corticoids systemic-therapy.
7. Known active infection including hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies).

   Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible.

   Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

   Subjects with HIV infection, and CD4+ T-cell (CD4+) counts < 350 cells/μL; or with acquired immunodeficiency syndrome (AIDS) - defining opportunistic infections within the past 12 months; or with uncontrolled opportunistic infections; or have an HIV viral load >400 copies/mL.
8. Subjects with uncontrollable severe active infections (such as septicemia, bacteremia, or viremia).
9. Subjects who received live attenuated vaccine within 4 weeks prior to the first dose of the investigational product, or plan to receive attenuated vaccine during the study.
10. Subjects who underwent a major surgery within 4 weeks prior to the first dose or plan to undergo a major surgery in 3 months after receiving the investigational drug (excluding catheterization, peripherally inserted central catheter, etc.).
11. Females who have a positive serum pregnancy test or who are lactating or planning to become pregnant during the study or within 6 months after the last dose of investigational product.
12. Received investigational therapy or used an investigational device within 4 weeks prior to the first dose of study treatment
13. History of psychiatric illness or substance abuse likely to interfere with the ability to comply with protocol requirements or giving informed consent
14. Prior malignancy active within the previous 3 years are not eligible for the trial except for: locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, prostate cancer with evidence of undetectable Prostate Specific Antigen (PSA) or carcinoma in situ of the prostate, cervix or breast.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-12-26 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
DLTs | Baseline up to 28 days after the first dose
  Dose Limiting Toxicities
MTD(maximum tolerated dose) | From start of treatment to treatment termination visit, up to 48 weeks
  To determine the maximum tolerated dose (MTD) of IMM47 in subjects with advanced solid tumors
adverse events (AEs) | Baseline up to 30 days after the last dose of study drug, up to 48 weeks
  Incidence and characteristics of adverse events (AEs)
RP2D (recommended Phase 2 dose) | From start of treatment to treatment termination visit, up to 48 weeks
  To determine the recommended Phase 2 dose (RP2D) of IMM47 in in subjects with advanced solid tumors
serious adverse events (SAEs) | Baseline up to 30 days after the last dose of study drug, up to 48 weeks
  Incidence and characteristics of serious adverse events (SAEs)

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 48 weeks of treatment cycles
  Maximum Plasma Concentration observed in patients with IMM47 dosed
Time to maximum concentration (Tmax) | 48 weeks of treatment cycles
  time to maximum concentration observed in patients with IMM47 dosed
Elimination half-life (t1/2) | 48 weeks of treatment cycles
  elimination half-life (t1/2) observed in patients with IMM47 dosed
Immunogenicity | 48 weeks of treatment cycles
  Positive rates of anti-drug antibodies (ADA)
Overall Rate Response (ORR) | When the last subject enrolled completes approximately 48 weeks of treatment
  ORR is defined as the proportion of participants who have a partial response (PR) or critical response (CR)
Disease control rate (DCR) | When the last subject enrolled completes approximately 48 weeks of treatment
  defined as the percentage of subjects with tumors who have complete response (CR), partial response (PR), and stable disease (SD)
Duration of response (DoR) | When the last subject enrolled completes approximately 48 weeks of treatment
  defined as the time from the first record of objective response to the first tumor progression or death of any cause
Progression-free Survival (PFS) | When the last subject enrolled completes approximately 48 weeks of treatment
  defined as the time from the start of treatment to tumor progression or death of any cause
AUC(0-tlast) | 48 weeks of treatment cycles
  area under the serum concentration-time curve from time 0 to the time of last quantifiable concentration (AUC0-tlast) in patients with IMM47 dosed
AUC0-inf | 48 weeks of treatment cycles
  area under the serum concentration-time curve from 0 to time infinity (AUC0-inf) in patients with IMM47 dosed

CONTACTS AND LOCATIONS:
Overall Officials: Jim Coward, A/Prof, Principal Investigator — Icon Cancer Centre South Brisbane, QLD; Charlotte Lemech, Dr, Principal Investigator — Scientia Clinical Research Ltd, NSW; Megan Crumbaker, Dr, Principal Investigator — Macquarie University Clinical Trials Unit (MQ CTU); David Martin, Dr, Principal Investigator — John Flynn Private Hospital, QLD
Locations (4):
- Australia (4):
  - Scientia Clinical Research Ltd, NSW, Sydney, New South Wales
  - Macquarie University Clinical Trials Unit (MQ CTU), Sydney, New South Wales
  - Icon Cancer Centre South Brisbane, QLD, Brisbane, Queensland
  - John Flynn Private Hospital, Gold Coast, Queensland

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: starting in Jun 1st 2025.